CLINICAL TRIAL: NCT04549597
Title: Randomized Open-Label Study to Evaluate Tenapanor as the Core Therapy in the Treatment of Hyperphosphatemia in Patients With Chronic Kidney Disease Who Are Phosphate Binder Naive or on Phosphate Binders to Optimize Phosphorus Management
Brief Title: Study to Evaluate the Use of Tenapanor as Core Therapy in the Treatment of Hyperphosphatemia
Acronym: OPTIMIZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEN-02-402
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Results first posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Hyperphosphatemia
Keywords: hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — tenapanor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Straight Switch (Experimental): Patients stop taking phosphate binders and start tenapanor 30 mg twice daily
  Interventions: Drug: Tenapanor
- Cohort 2: Decrease Phosphate Binder by 50% (Experimental): Decreases phosphate binder dose by at least 50% with the ability to switch the binder regiment from thrice daily (TID) to BID or once a day and initiates tenapanor 30 mg BID
  Interventions: Drug: Tenapanor
- Cohort 3: Phosphate Binder Naive (Experimental): Phosphate binder naive patients are enrolled as Cohort 3 and receive tenapanor with a starting dose of 30 mg/BID
  Interventions: Drug: Tenapanor

INTERVENTIONS:
Drug: Tenapanor — Use of tenapanor

SUMMARY:
This is a randomized, open-label study to evaluate different methods of initiating tenapanor therapy in CKD patients on dialysis with hyperphosphatemia, when they are either phosphate binder naïve or on phosphate binder therapy. The objective to evaluate the effect of tenapanor alone or in combination with phosphate binders to achieve target serum phosphorus (s-P) levels of ≤5.5 mg/dL when tenapanor is administered as the core therapy (alone or in combination with phosphate binders) for the treatment of hyperphosphatemia in patients with chronic kidney disease (CKD) on dialysis.

DETAILED DESCRIPTION:
Approximately 330 CKD patients on dialysis with hyperphosphatemia (>4.5 mg/dL) will be enrolled in this study.

This is a randomized, open-label study to evaluate different methods of initiating tenapanor therapy in CKD patients on dialysis with hyperphosphatemia, when they are either phosphate binder naïve or on phosphate binder therapy.

The study consists of a Screening visit and a 10-week open-label Treatment Period (TP), for which

* Patients with s-P >5.5 and ≤10.0 mg/dL under stable phosphate binder treatment are randomized in a 1:1 ratio to two different treatment cohorts:

  * Cohort 1 (straight switch), which stops taking phosphate binders and is started on tenapanor 30 mg twice daily (BID) at Visit 2 (Day 1);
  * Cohort 2, which decreases phosphate binder dose by at least 50% (may be more than 50% if patient is taking an odd number of binder pills each day), with ability to switch the binder regimen from thrice daily (TID) to BID or QD; and initiates tenapanor 30 mg BID at Visit 2 (Day 1).
* Phosphate binder naïve patients with s-P >4.5 and ≤10.0 mg/dL are enrolled as Cohort 3 and receive tenapanor at Visit 2 (Day 1) with a starting dose of 30 mg BID.
* Patients on phosphate binder therapy must receive phosphate binder(s) thrice daily, and both the s-P level assessed at the most recent measurement prior to the Screening visit (Visit 1) and the s-P level assessed at the Screening visit (Visit 1) must be >5.5 and ≤10.0 mg/dL to qualify for randomization into Cohort 1 or Cohort 2 at Visit 2 (Day 1).
* Phosphate binder naïve patients must have the s-P level assessed at the Screening visit (Visit 1) >4.5 and ≤10.0 mg/dL to qualify for enrollment into Cohort 3 at Visit 2 (Day 1).

Patients who do not meet the randomization/enrollment criteria on s-P will be discontinued as screen failures.

During the TP, patients will receive tenapanor starting at a dose of 30 mg twice daily. Tenapanor will be taken twice daily; just prior to breakfast and dinner. The Investigator may titrate the dose of tenapanor in 10 mg increments down to a minimum of 10 mg QD or up to a maximum of 30 mg BID at any time during the study based on s-P levels and/or gastrointestinal (GI) tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form prior to any study specific procedures.
2. Males or females aged 18 to 80 years, inclusive, at Screening (Visit 1).
3. Females must be non-pregnant and non-lactating.
4. Patients on phosphate binder therapy must be on chronic maintenance hemodialysis (HD) 3 times per week for at least 3 months or chronic maintenance peritoneal dialysis (PD) for a minimum of 6 months. If modality of dialysis has changed, the patient must meet one of the two dialysis criteria above and been on the new modality of dialysis for a minimum of one month. Phosphate binder naïve patients must be on chronic maintenance HD 3 times per week or chronic maintenance PD.
5. Kt/V ≥1.2 at most recent measurement prior to Screening (Visit 1).
6. Prescribed and taking phosphate binder medication at least 3 times per day or being phosphate binder naïve; defined as having not taken phosphate binders for at least 3 months prior to Screening. The patient must be taking a minimum of 6 pills per day for Renvela, Auryxia, or PhosLo; and/or a minimum of 3 pills per day for Fosrenol or Velphoro.
7. For patients taking phosphate binders, both the s-P level at the most recent measurement prior to Screening (Visit 1) and the s-P level at Screening (Visit 1) must be >5.5 and ≤10.0 mg/dL.
8. For phosphate binder naïve patients, the s-P level at Screening (Visit 1) must be >4.5 and ≤10.0 mg/dL.
9. Able to understand and comply with the protocol.

Exclusion Criteria:

1. Severe hyperphosphatemia defined as having an s-P level >10.0 mg/dL at any time point during routine clinical monitoring for the 3 preceding months before Screening (Visit 1).
2. Serum/plasma PTH >1200 pg/mL. The most recent value from the patient's medical records should be used.
3. Clinical signs of hypovolemia at Screening (Visit 1) as judged by the Investigator.
4. History of inflammatory bowel disease or irritable bowel syndrome with diarrhea.
5. Scheduled for living donor kidney transplant or plans to relocate to another center during the study.
6. Use of an investigational agent within 30 days prior to Screening (Visit 1).
7. Involvement in the planning and/or conduct of the study (applies to both Ardelyx/Contract Research Organization (CRO) staff and/or staff at the study site).
8. If, in the opinion of the Investigator, the patient is unable or unwilling to fulfill the requirements of the protocol or has a condition which would render the results uninterpretable.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- South Florida Research Institute, Lauderdale Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sprague SM, Weiner DE, Tietjen DP, Pergola PE, Fishbane S, Block GA, Silva AL, Fadem SZ, Lynn RI, Fadda G, Pagliaro L, Zhao S, Edelstein S, Spiegel DM, Rosenbaum DP. Tenapanor as Therapy for Hyperphosphatemia in Maintenance Dialysis Patients: Results from the OPTIMIZE Study. Kidney360. 2024 May 1;5(5):732-742. doi: 10.34067/KID.0000000000000387. Epub 2024 Feb 7. PMID 38323855
- [Derived] Silva AL, Chertow GM, Hernandez GT, Lynn RI, Tietjen DP, Rosenbaum DP, Yang Y, Edelstein S. Tenapanor Improves Long-Term Control of Hyperphosphatemia in Patients Receiving Maintenance Dialysis: the NORMALIZE Study. Kidney360. 2023 Nov 1;4(11):1580-1589. doi: 10.34067/KID.0000000000000280. Epub 2023 Oct 19. PMID 37853560

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Straight Switch): Patients stop taking phosphate binder and are immediately started on tenapanor 30 mg twice daily (BID)
- Cohort 2 (50% Phosphate Binder Reduction): Phosphate binder dose is decreased by at least 50% and tenapanor is initiated
Period: Overall Study
Arm/Group | Cohort 1 (Straight Switch) | Cohort 2 (50% Phosphate Binder Reduction) | Cohort 3: Phosphate Binder Naive
Started | 151 | 152 | 30
Completed | 127 | 133 | 25
Not Completed | 24 | 19 | 5

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Phosphate binders are stopped and tenapanor is started immediately upon enrollment
- Cohort 2: Phosphate binder dose is decreased by at least 50% and tenapanor is initiated
- Cohort 3: Phosphate Binder Naïve: Phosphate binder naive patients are enrolled as Cohort 3 and receive tenapanor with a starting dose of 30 mg/BID
  Tenapanor: Use of tenapanor
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3: Phosphate Binder Naïve | Total
Number analyzed (Participants) | 151 | 152 | 30 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.05) | 53.3 (12.16) | 55.4 (16.52) | 53.0 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 50 | 12 | 106
  Male | 107 | 102 | 18 | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 38 | 13 | 93
  Not Hispanic or Latino | 109 | 114 | 17 | 240
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 1 | 10
  Asian | 13 | 3 | 0 | 16
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 0 | 6
  Black or African American | 66 | 71 | 9 | 146
  White | 64 | 62 | 20 | 146
  More than one race | 2 | 4 | 0 | 6
  Unknown or Not Reported | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Effect of Tenapanor to Achieve Target s-P Levels of Less Than or Equal to 5.5 mg/dL
Description: To evaluate the effect of tenapanor alone or in combination with phosphate binders to achieve target serum phosphorus (s-P) levels of ≤5.5 mg/dL when tenapanor is administered as the core therapy for the treatment of hyperphosphatemia in patients with chronic kidney disease (CKD) on dialysis.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Straight Switch | Cohort 2: Decrease Phosphate Binder by 50% | Cohort 3: Phosphate Binder Naive
Number analyzed (Participants) | 151 | 152 | 30
Participants | 52 | 58 | 19

2. Secondary Outcome: To Evaluate the Effect of Tenapanor to Achieve Various s-P Levels ≤4.5 mg/dL
Description: Evaluating the ability of different treatment regimens to lower s-P to different levels
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Straight Switch | Cohort 2: Decrease Phosphate Binder by 50% | Cohort 3: Phosphate Binder Naive
Number analyzed (Participants) | 151 | 152 | 30
Participants | 18 | 23 | 13

3. Secondary Outcome: To Evaluate the Effect of Tenapanor on Reducing Daily Phosphorus-lowering Therapy Pill Burden.
Description: Evaluating the ability of tenapanor to make the phosphate lowering treatment regimen better for patients by evaluating the change in pill weight or pill number from baseline to the end of the 10-week treatment period.
Time Frame: 10 weeks
Population: Cohort 3 is not included since they are medication naive so there is no baseline pill weight
Measure: Median (Standard Deviation); unit: mg
Arm/Group | Cohort 1: Straight Switch | Cohort 2: Decrease Phosphate Binder by 50% | Cohort 3: Phosphate Binder Naive
Number analyzed (Participants) | 151 | 152 | 0
mg | -6262 (6149.7) | -3290 (5263.4) |

ADVERSE EVENTS:
Time Frame: 10 week treatment period followed by optional 16 week extension period
Groups:
- Cohort 1: Switch medication from phosphate binder to tenapanor upon enrollment
  Tenapanor: Use of tenapanor
- Cohort 2: Phosphate binder is decreased by at least 50% upon enrollment and tenapanor is added
  Tenapanor: Use of tenapanor
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3: Phosphate Binder Naïve
All-Cause Mortality (participants affected / at risk) | 1/151 | 1/152 | 0/30
Serious Adverse Events (participants affected / at risk) | 20/151 | 26/152 | 4/30
Other Adverse Events (participants affected / at risk) | 59/151 | 64/152 | 10/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=151) | Cohort 2 (N=152) | Cohort 3: Phosphate Binder Naïve (N=30)
Covid-19 (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Fluid Overload (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Arteriovenous Fistula Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=151) | Cohort 2 (N=152) | Cohort 3: Phosphate Binder Naïve (N=30)
Diarrhea (Gastrointestinal disorders) | 59 (59) | 64 (64) | 10 (10)

LIMITATIONS AND CAVEATS:
This was an open label study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications subject to the Sponsor's approval requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT04549597/Prot_SAP_000.pdf